CLINICAL TRIAL: NCT00521092
Title: Phase II Study of Sunitinib (SU11248) in Patients With Kaposi's Sarcoma in East Africa
Brief Title: Sunitinib Malate in Treating East African Patients With Kaposi Sarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00229; NCI-2009-00229 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 1706 - AMC 049; CDR0000561751; CASE 1706 / AMC 049 (Other: Case Comprehensive Cancer Center); 7831 (Other: CTEP); U01CA062502 (NIH); P30AI036219 (NIH)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2012-12

CONDITIONS: AIDS-related Kaposi Sarcoma; Classic Kaposi Sarcoma
Keywords: Treatment Experienced
MeSH Terms: conditions — AIDS-related Kaposi sarcoma | interventions — Sunitinib

ARMS (1):
- Arm I (Experimental): Patients receive oral sunitinib malate 50 mg once daily for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Procedure: laboratory biomarker analysis; Procedure: pharmacological study

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent
Procedure: laboratory biomarker analysis — Correlative study
Procedure: pharmacological study — Correlative study
  Other Names: pharmacological studies

SUMMARY:
Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. This phase II trial is studying the side effects and how well sunitinib malate works in treating patients with Kaposi sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the clinical response of sunitinib malate in patients with Kaposi sarcoma (KS) in Uganda and Kenya.

II. Compare clinical response rates in endemic versus epidemic (AIDS) KS. III. Determine the safety and tolerability of sunitinib malate in patients with endemic or epidemic (AIDS) KS.

SECONDARY OBJECTIVES:

I Monitor the impact of sunitinib malate on underlying HIV-1 and Kaposi sarcoma-associated herpesvirus (KSHV) viral infection (HIV-1 plasma RNA and KSHV cell-associated DNA).

II. Evaluate morphological changes in KS lesions after treatment. III. Determine the pharmacokinetic profile of sunitinib malate in patients with KS.

IV Evaluate KSHV gene expression in endemic and epidemic KS lesions in patients in Uganda and Kenya.

OUTLINE: This is a multicenter study. Patients are stratified according to HIV-serostatus (endemic [HIV-seronegative] vs epidemic [HIV-seropositive/AIDS] kaposi sarcoma).

Patients receive oral sunitinib malate 50 mg once daily for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection periodically for correlative and pharmacokinetic studies. Samples are analyzed for CD4 lymphocyte counts, HIV-1 plasma RNA levels, KSHV specific antibodies, expression pattern of KSHV in vitro and in vivo, expression of latently versus lytically expressed genes in tumor tissue, and plasma concentrations of sunitinib malate and its active metabolite, SU12662.

After completion of study treatment, patients are followed every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-1
* Documented HIV-serostatus [HIV-seronegative (endemic KS) or HIV-seropositive (epidemic/AIDS KS)]
* No symptomatic organ involvement, visceral crisis, or life-threatening disease (e.g., extensive or symptomatic pulmonary disease or reticuloendothelial system/hepatic involvement) for which aggressive double- or triple-drug combination chemotherapy for urgent cytoreduction is indicated (i.e., doxorubicin hydrochloride, bleomycin, and vinblastine [ABV], BV, or AV)
* Histologically confirmed Kaposi sarcoma
* Platelet count > 75,000/uL
* Life expectancy >= 24 weeks
* Absolute granulocyte count > 1,000/uL
* Hemoglobin > 8.0 g/dL OR hematocrit > 24%
* Serum creatinine =< 2.0 mg/dL
* AST < 3 times normal
* Fertile patients must use effective contraception
* Normal clinical cardiac examination and normotensive (systolic and diastolic BP < 140/90 mm Hg) documented on at least two occasions prior to enrollment
* Normal ECG including QTc interval < 500 msec
* Normal echocardiogram prior to enrollment (if feasibly possible)
* Must be able to swallow study medication
* No acute infections [Patients with chronic infections (e.g., malaria, tuberculosis, parasitic infections, or hepatitis B or C) that may be active but under treatment are allowed provided all eligibility criteria are met]
* At least 60 days since prior local treatment modalities (e.g., resection, cryosurgery, radiotherapy, or intralesional therapy) AND treated lesions must have clearly progressed following such therapies if the lesions are to be used as an index lesion
* No prior systemic anticancer therapy for Kaposi sarcoma
* Concurrent antiretroviral therapy required for HIV-seropositive patients (Patient must be on a stable regimen 8 weeks prior to study enrollment--An exception may be made for patients who have exhausted or are intolerant to all available regimens)
* No other concurrent systemic anticancer therapy
* Patient resides in Uganda or Kenya, East Africa

Exclusion Criteria:

* Pregnant or nursing
* Baseline diarrhea >= grade 2 by CTCAE
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or acute active infection
  * Symptomatic congestive heart failure (NYHA class III or IV heart disease)
  * Unstable angina pectoris
* Uncontrolled intercurrent illness including, but not limited to, any of the following: 1) Cardiac arrhythmia (i.e., history of serious ventricular arrhythmia, ventricular fibrillation, or ventricular tachycardia >= 3 beats in a row OR QTc >= 500 msec) 2) Psychiatric illness or social situation that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 11 months
  The true response rate will be estimated based on the number of responses using a binomial distribution. The confidence intervals for them can be estimated using same distribution. Chi-square test or Fisher's exact test will be used to examine the difference of response rate between the two cohorts and log-rank test for the difference of survival outcomes.
Overall survival | From the date of treatment to date of death, assessed up to 11 months
  Will be estimated by Kaplan-Meier method.
Progression-free survival | From the date of treatment to date of death or date of disease progression, assessed up to 11 months
  Will be estimated by Kaplan-Meier method.
Levels of plasma-associated HIV-1 RNA viral load and cell-associated KSHV DNA viral load | Up to 11 months
  Multivariate analysis will be performed using the Cox proportional hazards model. The effects of CD4+ lymphocyte counts, plasma HIV-1 RNA viral load and KSHV DNA level on the objective response rate will be evaluated using multivariate logistic regression.

SECONDARY OUTCOMES:
Changes in CD4+ and CD8+ cell counts, levels of plasma-associated HIV-1 RNA, and cell-associated KSHV DNA load | Baseline and 6 weeks
  For each treatment cohort and for all groups combined, the Wilcoxon signed rank test (the non-parametric version of paired T-test) will be used to evaluate the changes.

CONTACTS AND LOCATIONS:
Overall Officials: Scot Remick, Principal Investigator — Case Comprehensive Cancer Center